CLINICAL TRIAL: NCT01806259
Title: Perioperative Ketorolac in High Risk Breast Cancer Patients With and Without Inflammation. A Prospective Randomized Placebo-controlled Trial.
Brief Title: Ketorolac in Breast Cancer Surgery
Acronym: KBCt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Anticancer Fund, Belgium (Other)
Responsible Party: Principal Investigator, Patrice Forget, Docteur, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBCtrial
Record Dates: First submitted 2013-02-20; First posted 2013-03-07 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Curative Breast Cancer Surgery; Inflammatory Positive/Negative Status; Pre Surgical Incision Administration
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ketorolac 30 mg (Experimental): Active drug to be compared with placebo
  Interventions: Drug: Ketorolac 30 mg IV
- NaCl 0.9% 3mL (Placebo Comparator): Placebo looking like the Active drug
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ketorolac 30 mg IV — Active drug
  Other Names: ketorolac tromethamine
  Arms: ketorolac 30 mg
Drug: Placebos — Placebo looking like the Active drug
  Other Names: NaCl 0.9%
  Arms: NaCl 0.9% 3mL

SUMMARY:
Do the use of Ketorolac in one intravenous injection at the moment of the operative incision reduce the number of recurrence in patient with advanced breast cancer without inflammation signs.

ELIGIBILITY:
Inclusion Criteria:

Written informed Consent age : 18-85 years weight: 50-100 kg Neutrophils / Lymphocytes ratio >4 and/or "triple negative" histological status and/or Positive lymph nodes

Exclusion Criteria:

Previous cancer (behalf of basocellular skin cancer and in situ uterine cervix cancer) Non compliance or refusal of the protocol Positive Pregnancy test Childbearing or breastfeeding mothers Contra-indication for NSAIDs NSAIDs intake in the 5 days before randomisation NSAIDs use planned in the 30 days after randomisation Non curative surgery (T4 or M1 tumor classification )

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Forget, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Background] Forget P, Vandenhende J, Berliere M, Machiels JP, Nussbaum B, Legrand C, De Kock M. Do intraoperative analgesics influence breast cancer recurrence after mastectomy? A retrospective analysis. Anesth Analg. 2010 Jun 1;110(6):1630-5. doi: 10.1213/ANE.0b013e3181d2ad07. Epub 2010 Apr 30. PMID 20435950
- [Derived] Forget P, Bouche G, Duhoux FP, Coulie PG, Decloedt J, Dekleermaker A, Guillaume JE, Ledent M, Machiels JP, Mustin V, Swinnen W, van Maanen A, Vander Essen L, Verougstraete JC, De Kock M, Berliere M. Intraoperative ketorolac in high-risk breast cancer patients. A prospective, randomized, placebo-controlled clinical trial. PLoS One. 2019 Dec 4;14(12):e0225748. doi: 10.1371/journal.pone.0225748. eCollection 2019. PMID 31800611
- [Derived] Forget P, Berliere M, van Maanen A, Duhoux FP, Machiels JP, Coulie PG, Bouche G, De Kock M; Ketorolac in Breast Cancer trial (KBCtrial) group. Perioperative ketorolac in high risk breast cancer patients. Rationale, feasibility and methodology of a prospective randomized placebo-controlled trial. Med Hypotheses. 2013 Oct;81(4):707-12. doi: 10.1016/j.mehy.2013.07.033. Epub 2013 Aug 9. PMID 23937996
- See also: Related Info — http://www.anesthesia-analgesia.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac 30 mg: Active drug to be compared with placebo
  Ketorolac 30 mg IV
- NaCl 0.9% 3mL: Placebo
Period: Overall Study
Arm/Group | Ketorolac 30 mg | NaCl 0.9% 3mL
Started | 96 | 107
Completed | 96 | 107
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NaCl 0.9% 3mL: Ketorolac 30 mg IV
- Total: Total of all reporting groups
Arm/Group | Ketorolac 30 mg | NaCl 0.9% 3mL | Total
Number analyzed (Participants) | 96 | 107 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (14) | 55.4 (13.9) | 55.7 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 107 | 202
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival
Description: 2 years for the primary analysis + 3 additional years for secondary analysis (From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years)
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac 30 mg | NaCl 0.9% 3mL
Number analyzed (Participants) | 96 | 107
Participants | 80 | 96

2. Other Pre Specified Outcome: Overall Survival
Description: 2 years for the primary analysis + 3 additional years for secondary analysis (From date of randomization until the date of death from any cause assessed up to 5 years)
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac 30 mg | NaCl 0.9% 3mL
Number analyzed (Participants) | 96 | 107
Participants | 93 | 105

ADVERSE EVENTS:
Arm/Group | Ketorolac 30 mg | NaCl 0.9% 3mL
Serious Adverse Events (participants affected / at risk) | 8/96 | 7/107
Other Adverse Events (participants affected / at risk) | 0/96 | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac 30 mg (N=96) | NaCl 0.9% 3mL (N=107)
Any type (not bleeding related) (General disorders) | 7 (7) | 7 (7)
Hematoma requiring surgery (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes